CLINICAL TRIAL: NCT04515173
Title: Artificial Intelligence for Enhancing the Diagnosis and Treatment of Mental Illness：a Prospective, Randomized Controlled Multicenter Clinical Trail
Brief Title: Artificial Intelligence in Mental Illness Diagnosis and Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Yifeng XU, The director of the hospital, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: "Six zero zero"robot
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Artificial Intelligence; Mental Illness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial intelligence group (Experimental): On the basis of conventional drug therapy combined with psychotherapy robot psychotherapy, the corresponding intelligent psychotherapy module and intensity were recommended according to the results of intelligent psychological evaluation. Each module was set once a week, 50 minutes each time, a total of 12 times.
  Interventions: Diagnostic Test: Artificial intelligence diagnosis and treatment assistance system
- General group (Other): The subjects in this group only received routine drug therapy and routine outpatient follow-up evaluation
  Interventions: Diagnostic Test: Artificial intelligence diagnosis and treatment assistance system

INTERVENTIONS:
Diagnostic Test: Artificial intelligence diagnosis and treatment assistance system — An artificial intelligence robot that can assist psychiatrists in disease screening, diagnosis, treatment, and follow-up.

SUMMARY:
To improve the quality of mental health services, we will develop a robot that includes disease screening, diagnosis, treatment, and follow-up. The effectiveness of robots will be verified in a prospective, randomized, multi-center clinical trial. We assume that the robot will reduce the differences in the experience of doctors of different years and will improve mental health care across the country, and improve the uneven distribution of mental health resources through remote resource sharing.

DETAILED DESCRIPTION:
Anxiety disorder is the most common mental disorder in the world. The lifetime prevalence of anxiety disorder in China is as high as 7.6%, but the treatment rate is less than 30%, and the standard treatment rate is only 9.8%. The disease burden is heavy, and it is one of the most serious public health problems in China. Anxiety disorder is a chronic relapsing disease, single drug treatment only 35-50% efficient, psychological treatment as the most international evidence-based foundation and anxiety disorder most commonly used treatment method, can be a single treatment for anxiety disorders or improve the effect of the medication, but because of clinical psychology in China started late, the lack of professionals, unable to meet the huge demand for psychological treatment in our country, therefore, how to develop efficient and standardized anxiety disorders psychotherapy pattern, improve the psychological treatment of acquired, is the key to improve the clinical curative effect of anxiety disorders. Based on the intelligent assisted psychotherapy system based on cognitive behavior and mindfulness developed in the early stage, this research group established the accurate psychotherapy artificial intelligence robot based on evaluation to assist the whole process of standardized psychotherapy for anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* Community high-risk groups and institutional groups.
* According to the ICD-11 diagnostic guidelines of anxiety-related disorders, depression-related disorders, addiction-related disorders, compulsive-related disorders diagnosis,
* age 18-60 years old,
* skilled in the operation of computers or smartphones,
* language, reading ability is normal,
* willing to participate in the project and sign informed consent study.

Exclusion Criteria:

* The symptoms of mental illness are severe and require hospitalization, or the patient is unable to complete the required assessment examination and treatment.
* Those who have a higher risk of self-injury or suicide.
* People with severe physical illness, central system disease, or substance abuse.
* Receive physical therapy at the same time.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4000 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
System sensitivity | Baseline
  The proportion that the system correctly determines people who are actually sick to be true.
System specificity | Baseline
  The proportion that the system correctly determines people who are actually disease-free to be true negative.
Cure rate | 24 weeks
  End of the period reached the total number of clinically cured patients / total number of all patients involved in the study
Recurrence rate | 24 weeks
  Total number of patients with recurrence or recurrence of symptoms/total number of patients involved in the study

SECONDARY OUTCOMES:
Patients' satisfaction | Baseline, 12 weeks, 24 weeks
  The degree of patient satisfaction with the system
Clinical global impressions | Baseline, 12 weeks, 24 weeks
  The score of clinical global impressions scale(CGI)
Social function | Baseline, 12 weeks, 24 weeks
  The score of social disability screening schedule(SDSS）
Doctors' satisfaction | Baseline, 12 weeks, 24 weeks
  The degree of doctors' satisfaction with the system

CONTACTS AND LOCATIONS:
Overall Officials: Yifeng Xu, Study Chair — SMHC; Jianyin QIU, Study Director — SMHC